CLINICAL TRIAL: NCT01017523
Title: Improving Diabetes Outcome: The Diabetes Support Project
Brief Title: Diabetes Support Project: Couples Intervention
Acronym: DSP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paula Trief, Professor of Psychiatry and Medicine, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5840; R18DK080867 (NIH)
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; relationship; social support; telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Couples) (Experimental): Diabetes self-management education, telephone support and behavior change for couples.
  Interventions: Behavioral: Telephone support and behavior change
- 2 (Individual) (Active Comparator): Diabetes self-management education, telephone support and behavior change for individuals.
  Interventions: Behavioral: Telephone support and behavior change
- 3 (Control) (Placebo Comparator): Diabetes self-management education only.
  Interventions: Other: Diabetes self-management education

INTERVENTIONS:
Behavioral: Telephone support and behavior change — Diabetes self-management education provided over the telephone either for individual or couples
  Arms: 1 (Couples); 2 (Individual)
Other: Diabetes self-management education — Limited diabetes self-management education provided over the telephone, serves as an enhanced usual care control intervention
  Arms: 3 (Control)

SUMMARY:
Research has shown that diabetes affects both the patient and family, and that support from family and partners helps diabetes patients manage their illness better. However, diabetes programs rarely involve the partner. The purpose of this study is to test an intervention that helps partners and patients who have type 2 diabetes better support each other. The intervention will be delivered over the telephone to reach more people. Our hypothesis is that an intervention that targets the couple has a greater effect on health and well-being of patients than one that targets the individual patient alone.

DETAILED DESCRIPTION:
Diabetes is a serious illness that affects an estimated 7% of the US population, and is associated with life-threatening and disabling complications. Research has shown that diabetes affects both the patient and family, and that support from one's spouse has been found to be the most important source of support during illness episodes. Research clearly shows that marital interaction, i.e., how the support is given and received, impacts both marital quality and health functioning. Despite the acknowledged importance of social support, the vast majority of chronic illness interventions target the individual patient. Telephone counseling has been effectively used to enhance feasibility and target patients with many illnesses, and has many benefits including low cost, decreased subject burden, and the ability to reach a broader population. This study proposes a study of a telephone-administered behavior change that promotes couples communication and collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* A1c level is >=7.5%
* Age of target subject and spouse/partner is 21 years or older
* Married or together for > 1 year
* Able to speak, read, and hear English
* Have a telephone

Exclusion Criteria:

* History of diabetes-related medical complications
* History of active psychosis or dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose control (hemoglobin AIc) | Baseline, and 3 follow ups (mos 4, 8, 12)

SECONDARY OUTCOMES:
BMI/Waist circumference | Baseline and 3 follow-ups (mos 4, 8, and 12)
Measures of behavior change (diet, physical activity) | Baseline and 3 follow-ups (mos 4, 8, and 12)
Diabetes-related quality of life outcome (distress) | Baseline and 3 follow-ups (mos 4, 8, and 12)

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Trief, Ph.D., Principal Investigator — State University of New York - Upstate Medical University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - SUNY Upstate Medical University, Dept. of Psychiatry, Syracuse, New York

REFERENCES:
- [Background] Fisher L, Chesla CA, Bartz RJ, Gilliss C, Skaff MA, Sabogal F, Kanter RA, Lutz CP. The family and type 2 diabetes: a framework for intervention. Diabetes Educ. 1998 Sep-Oct;24(5):599-607. doi: 10.1177/014572179802400504. PMID 9830956
- [Background] Fisher L, Weihs KL. Can addressing family relationships improve outcomes in chronic disease? Report of the National Working Group on Family-Based Interventions in Chronic Disease. J Fam Pract. 2000 Jun;49(6):561-6. PMID 10923558
- [Background] Trief PM, Grant W, Elbert K, Weinstock RS. Family environment, glycemic control, and the psychosocial adaptation of adults with diabetes. Diabetes Care. 1998 Feb;21(2):241-5. doi: 10.2337/diacare.21.2.241. PMID 9539989
- [Background] Trief PM, Ploutz-Snyder R, Britton KD, Weinstock RS. The relationship between marital quality and adherence to the diabetes care regimen. Ann Behav Med. 2004 Jun;27(3):148-54. doi: 10.1207/s15324796abm2703_2. PMID 15184090
- [Background] Trief PM, Himes CL, Orendorff R, Weinstock RS. The marital relationship and psychosocial adaptation and glycemic control of individuals with diabetes. Diabetes Care. 2001 Aug;24(8):1384-9. doi: 10.2337/diacare.24.8.1384. PMID 11473074
- [Background] Trief PM, Wade MJ, Britton KD, Weinstock RS. A prospective analysis of marital relationship factors and quality of life in diabetes. Diabetes Care. 2002 Jul;25(7):1154-8. doi: 10.2337/diacare.25.7.1154. PMID 12087013
- [Background] Garfield SA, Malozowski S, Chin MH, Narayan KM, Glasgow RE, Green LW, Hiss RG, Krumholz HM; Diabetes Mellitus Interagency Coordinating Committee (DIMCC) Translation Conference Working Group. Considerations for diabetes translational research in real-world settings. Diabetes Care. 2003 Sep;26(9):2670-4. doi: 10.2337/diacare.26.9.2670. No abstract available. PMID 12941736
- [Background] Delamater AM, Jacobson AM, Anderson B, Cox D, Fisher L, Lustman P, Rubin R, Wysocki T; Psychosocial Therapies Working Group. Psychosocial therapies in diabetes: report of the Psychosocial Therapies Working Group. Diabetes Care. 2001 Jul;24(7):1286-92. doi: 10.2337/diacare.24.7.1286. PMID 11423517
- [Background] Kiecolt-Glaser JK, Newton TL. Marriage and health: his and hers. Psychol Bull. 2001 Jul;127(4):472-503. doi: 10.1037/0033-2909.127.4.472. PMID 11439708
- [Derived] Yorgason JB, Sandberg JG, Weinstock RS, Trief PM, Fisher L, Hessler D. The importance of relationship processes for lowering BMI over time in women with type 2 diabetes in a randomized controlled trial. Obes Res Clin Pract. 2019 Nov-Dec;13(6):599-601. doi: 10.1016/j.orcp.2019.08.003. Epub 2019 Oct 22. PMID 31653476
- [Derived] Trief PM, Fisher L, Sandberg J, Hessler DM, Cibula DA, Weinstock RS. Two for one? Effects of a couples intervention on partners of persons with Type 2 diabetes: a randomized controlled trial. Diabet Med. 2019 Apr;36(4):473-481. doi: 10.1111/dme.13871. Epub 2019 Jan 8. PMID 30485516
- [Derived] Trief PM, Fisher L, Sandberg J, Cibula DA, Dimmock J, Hessler DM, Forken P, Weinstock RS. Health and Psychosocial Outcomes of a Telephonic Couples Behavior Change Intervention in Patients With Poorly Controlled Type 2 Diabetes: A Randomized Clinical Trial. Diabetes Care. 2016 Dec;39(12):2165-2173. doi: 10.2337/dc16-0035. Epub 2016 Jul 25. PMID 27456837